CLINICAL TRIAL: NCT01106157
Title: Reversing Type 1 Diabetes After it is Established: A Pilot Safety and Feasibility Study of Anti-Thymocyte Globulin (Thymoglobulin®)and Pegylated GCSF (Neulasta®) in Established Type 1 Diabetes
Brief Title: Reversing Type 1 Diabetes After it is Established
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UF-ATG-GCSF001; IRB201702525 (Other: University of Florida); 041-2010 (Other: Univeristy of Florida); OCR16038 (Other: University of Florida)
Record Dates: First submitted 2010-04-15; First posted 2010-04-19 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Autoimmune, Diabetes Mellitus, Glucose Metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — thymoglobulin; pegfilgrastim

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anti-Thymocyte Globin plus pegylated GCSF (Experimental): Subjects will receive an infusion of Anti-Thymocyte Globin (ATG) followed by 6 doses of pegylated GCSF every 2 weeks for 10 weeks.
  Interventions: Drug: Anti-Thymocyte Globin (ATG); Drug: Pegylated GCSF
- Placebo (Placebo Comparator): Saline infusion will be given on both Day 1 and Day 2 followed by placebo injection given in identical volumes in identical syringes in the identical subcutaneous manner
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anti-Thymocyte Globin (ATG) — Anti-Thymocyte Globin (ATG) will be given as 0.5/mg/kg on day 1 and 2mg/kg on day 2.
  Other Names: Thymoglobulin
  Arms: Anti-Thymocyte Globin plus pegylated GCSF
Drug: Placebo — Saline infusions will be given on Day 1 and Day 2 followed by placebo injections given in identical volumes in identical syringes
  Other Names: Saline infusion
  Arms: Placebo
Drug: Pegylated GCSF — 6 doses of pegylated GCSF (6mg/dose) will be given subcutaneously every 2 weeks beginning after the ATG infusion.
  Other Names: Neulasta
  Arms: Anti-Thymocyte Globin plus pegylated GCSF

SUMMARY:
The primary purpose of this study is to determine if giving the combination therapy consisting of Thymoglobulin® (ATG) and Neulasta® (GCSF) to patients with established Type 1 Diabetes (T1D) is safe and secondarily, if the ATG and GCSF will preserve insulin production.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, phase I/II trial. Potential subjects will be screened via a 4 hour mixed meal tolerance test to assess residual beta cell (C-peptide) function. If the C-peptide level at any time is ≥ 0.1 pmol/ml, and the subject meets the additional inclusion and exclusion criteria, they will be eligible for randomization and enrollment. The study will be randomized 2:1 such that 17 subjects will receive active therapy and 8 will receive placebo. Subjects must receive Thymoglobulin®/ Neulasta® or placebo within 8 weeks of randomization. Thymoglobulin® (2.5mg/kg)/placebo will be given as 0.5 mg/kg IV on day 1 and 2 mg/kg on day 2. Six doses of Neulasta® (6mg/dose)/placebo will be given as standard of care every 2 weeks, with the first dose given prior to discharge after the Thymoglobulin® infusion. Complete metabolic panel (CMP) and complete blood count (CBC) will be done at the screening visit, just prior to study drug initiation, daily during the Thymoglobulin® infusion admission, and at follow up visits. Following discharge, daily phone calls will be made to the subjects during the first 5 days of therapy and weekly thereafter. In addition, weekly phone calls for the month following completion of therapy will be used to document adverse reactions. Thereafter calls will be made every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must be > 12 years < 45
* Must have a diagnosis of T1D of greater than 4 months duration, with an upper limit of 2 years, Now only recruiting for those diagnosed greater than 1 year but less than 2 years.
* Must have at least one diabetes-related autoantibody present (e.g., islet cell autoantigen (ICA), GAD, ZnT8, or islet antigen 2 (IA2) autoantibodies)
* Must have stimulated C-peptide levels ≥ 0.1 pmol/ml (0.3ng/mL) when measured during a mixed meal tolerance test (MMTT), conducted at least 4 months from diagnosis of diabetes, and within 8 weeks of randomization
* Must be EBV PCR negative within two weeks of randomization if EBV seronegative at screening
* Be at least 6 weeks from last live immunization
* Be willing to forgo live vaccines for 3 months following last dose of study drug
* Be willing to comply with intensive diabetes management
* Normal screening values for complete blood count (CBC), renal function and electrolytes (CMP).

Exclusion Criteria:

* Be immunodeficient or have clinically significant chronic lymphopenia: (Leukopenia (< 3,000 leukocytes /μL), neutropenia (<1,500 neutrophils/μL), lymphopenia (<800 lymphocytes/μL), or thrombocytopenia (<125,000 platelets/μL).
* Have a chronic infection at time of randomization
* Have a positive PPD
* Be currently pregnant or lactating, or anticipate getting pregnant within the next two years
* Require use of other immunosuppressive agents
* Have serologic evidence of current or past HIV, Tuberculosis, Hepatitis B or Hepatitis C infection
* Have any complicating medical issues or abnormal clinical laboratory results that interfere with study conduct, or cause increased risk to include pre-existing cardiac disease, chronic obstructive pulmonary disease (COPD), sickle cell disease, neurological, or blood count abnormalities (e.g., lymphopenia, leukopenia, or thrombocytopenia)
* Have a history of malignancies
* Evidence of liver dysfunction with angiotensin sensitivity test (AST) or ALT greater than 3 times the upper limits of normal
* Evidence of renal dysfunction with creatinine greater than 1.5 times the upper limit of normal
* Vaccination with a live virus within the last 6 weeks
* Current use of non-insulin pharmaceuticals that affect glycemic control
* Active participation in another T1D treatment study in the previous 30 days
* Known allergy to G-CSF or ATG
* Prior treatment with ATG or known allergy to rabbit derived products
* Any condition that in the investigator's opinion, may adversely affect study participation or may compromise the study results

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Haller, MD, Principal Investigator — University of Florida Pediatric Endocrinology
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - University of Florida, Gainesville, Florida

REFERENCES:
- [Background] Parker MJ, Xue S, Alexander JJ, Wasserfall CH, Campbell-Thompson ML, Battaglia M, Gregori S, Mathews CE, Song S, Troutt M, Eisenbeis S, Williams J, Schatz DA, Haller MJ, Atkinson MA. Immune depletion with cellular mobilization imparts immunoregulation and reverses autoimmune diabetes in nonobese diabetic mice. Diabetes. 2009 Oct;58(10):2277-84. doi: 10.2337/db09-0557. Epub 2009 Jul 23. PMID 19628781
- [Derived] Haller MJ, Gitelman SE, Gottlieb PA, Michels AW, Rosenthal SM, Shuster JJ, Zou B, Brusko TM, Hulme MA, Wasserfall CH, Mathews CE, Atkinson MA, Schatz DA. Anti-thymocyte globulin/G-CSF treatment preserves beta cell function in patients with established type 1 diabetes. J Clin Invest. 2015 Jan;125(1):448-55. doi: 10.1172/JCI78492. Epub 2014 Dec 15. PMID 25500887
- See also: University of Florida Diabetes Center of Excellence — http://diabetes.ufl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Anti-Thymocyte Globin Plus Pegylated GCSF: Subjects will receive an infusion of Anti-Thymocyte Globin (ATG) followed by 6 doses of pegylated GCSF every 2 weeks for 10 weeks.
  Anti-Thymocyte Globin plus pegylated GCSF: Anti-Thymocyte Globin (ATG)will be given as 0.5/mg/kg on day 1 and 2mg/kg on day 2, plus 6 doses of pegylated GCSF (6mg/dose) given subcutaneously every 2 weeks beginning after the ATG infusion.
Period: Overall Study
Arm/Group | Anti-Thymocyte Globin Plus Pegylated GCSF | Placebo
Started | 17 | 8
Completed | 16 | 8
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Anti-Thymocyte Globin Plus Pegylated GCSF: Subjects will receive an infusion of Anti-Thymocyte Globin (ATG) followed by 6 doses of pegylated GCSF every 2 weeks for 10 weeks.
  Anti-Thymocyte Globin plus pegylated GCSF: Anti-Thymocyte Globin (ATG)will be given as 0.5/mg/kg on day 1 and 2mg/kg on day 2, plus 6 doses of pegylated GCSF (6mg/dose)given subcutaneously every 2 weeks beginning after the ATG infusion
- Total: Total of all reporting groups
Arm/Group | Anti-Thymocyte Globin Plus Pegylated GCSF | Placebo | Total
Number analyzed (Participants) | 17 | 8 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 5 | 10
  Between 18 and 65 years | 12 | 3 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.64 (10) | 23.55 (10.6) | 23.61 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 12 | 5 | 17
Region of Enrollment [Number; unit: participants]
  United States | 17 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Metabolic Function Baseline to 12 Months.
Description: Area Under Curve (AUC) C-peptide production. Subjects underwent a 2 hour mixed meal tolerance test (MMTT) using a 6ml/kg load of boost to stimulate insulin production. Samples were collected at baseline, 10 minutes, 20 minutes, 30 minutes, 60 minutes, 90 minutes, and 120 minutes. AUC was then calculated. Subjects repeated the MMTT at baseline, 3, 6, 9, and 12 months following ATG/GCSF or placebo. The primary outcome for the study was the change over 12 months in AUC C-peptide (1 year - baseline) for those who received ATG/GCSF versus the change in AUC C-peptide (1 year - baseline) for those who received placebo
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: nmol/L/min
Arm/Group | Anti-Thymocyte Globin Plus Pegylated GCSF | Placebo
Number analyzed (Participants) | 16 | 8
nmol/L/min | 0.74 (0.47) | 0.43 (0.32)
Statistical Analysis 1: Comparison: Anti-Thymocyte Globin Plus Pegylated GCSF vs Placebo; Test type: Superiority or Other; p = 0.017, t-test, 2 sided; Mean Difference (Net) = 0.277, 95% CI 2-sided [0.001 to 0.552], Standard Error of Mean 0.134

2. Secondary Outcome: Percent Change in Regulatory T Cells (Treg) Baseline to 12 Months
Description: Change in regulatory T cells (Treg) baseline to 12 months
Time Frame: Change in Baseline to 12 months
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Anti-Thymocyte Globin Plus Pegylated GCSF | Placebo
Number analyzed (Participants) | 16 | 8
percentage change | -0.46 (0.36) | 0 (.036)
Statistical Analysis 1: Comparison: Anti-Thymocyte Globin Plus Pegylated GCSF vs Placebo; Test type: Superiority or Other; p = 0.43, t-test, 2 sided; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.30 to 0.13], Standard Error of Mean 0.104

3. Secondary Outcome: A1c
Description: Change in A1c baseline to 12 months
Time Frame: Change in baseline to 12 months
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Anti-Thymocyte Globin Plus Pegylated GCSF | Placebo
Number analyzed (Participants) | 16 | 8
% change | 0.47 (1.88) | 0.98 (0.79)
Statistical Analysis 1: Comparison: Anti-Thymocyte Globin Plus Pegylated GCSF vs Placebo; Test type: Superiority or Other; p = 0.37, t-test, 2 sided; Mean Difference (Net) = -0.51, 95% CI 2-sided [-1.64 to 0.63], Standard Error of Mean 0.70

4. Secondary Outcome: Change in Insulin Requirements, Baseline to 12 Months
Description: Change in Insulin Requirements, baseline to 12 months
Time Frame: Change from baseline to 12 months
Population: Insulin use data was not provided by all subjects resulting in sampling for analysis that was smaller than the cohort for the entire study.
Measure: Mean (Standard Deviation); unit: units/kg/day
Arm/Group | Anti-Thymocyte Globin Plus Pegylated GCSF | Placebo
Number analyzed (Participants) | 14 | 5
units/kg/day | -0.03 (0.4) | 0.08 (0.19)
Statistical Analysis 1: Comparison: Anti-Thymocyte Globin Plus Pegylated GCSF vs Placebo; Test type: Superiority or Other; p = 0.69, t-test, 2 sided; Mean Difference (Net) = -0.064, 95% CI 2-sided [-0.40 to 0.27], Standard Error of Mean 0.16

5. Secondary Outcome: Change in Glutamic Acid Decarboxylase Antibodies (GADA) From Baseline to 12 Months
Description: Change in Glutamic Acid Decarboxylase Antibodies (GADA) over 12 months
Time Frame: Change from baseline to 12 months
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Anti-Thymocyte Globin Plus Pegylated GCSF | Placebo
Number analyzed (Participants) | 16 | 8
nmol/L | -17.75 (225.81) | -29.5 (38.96)
Statistical Analysis 1: Comparison: Anti-Thymocyte Globin Plus Pegylated GCSF vs Placebo; Test type: Superiority or Other; p = 0.89, t-test, 2 sided; Mean Difference (Net) = 11.75, 95% CI 2-sided [-156.8 to 180.3], Standard Error of Mean 81.3

6. Secondary Outcome: Change in Insulin Autoantibodies (IAA) From Baseline to 12 Months
Description: Change in Insulin Autoantibodies (IAA) over 12 months
Time Frame: Change from baseline to 12 months
Measure: Mean (Standard Deviation); unit: Units/mL
Arm/Group | Anti-Thymocyte Globin Plus Pegylated GCSF | Placebo
Number analyzed (Participants) | 16 | 8
Units/mL | 0.12 (0.5) | -0.15 (0.43)
Statistical Analysis 1: Comparison: Anti-Thymocyte Globin Plus Pegylated GCSF vs Placebo; Test type: Superiority or Other; p = 0.2, t-test, 2 sided; Mean Difference (Net) = 0.28, 95% CI 2-sided [-0.15 to 0.70], Standard Error of Mean 0.21

7. Secondary Outcome: Change in Insulinoma Associated 2 Autoantibodies (IA-2A) From Baseline to 12 Months
Description: Change in Insulinoma Associated 2 Autoantibodies (IA-2A)
Time Frame: Change from baseline to 12 months
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Anti-Thymocyte Globin Plus Pegylated GCSF | Placebo
Number analyzed (Participants) | 16 | 8
nmol/L | -21.63 (50.3) | 2.5 (31.47)
Statistical Analysis 1: Comparison: Anti-Thymocyte Globin Plus Pegylated GCSF vs Placebo; Test type: Superiority or Other; p = 0.23, t-test, 2 sided; Mean Difference (Net) = -24.13, 95% CI 2-sided [-64.8 to 16.7], Standard Error of Mean 19.61

8. Secondary Outcome: Change in Zinc Transporter 8 Autoantibodies (ZnT8A) From Baseline to 12 Months
Description: Change in Zinc Transporter 8 Autoantibodies (ZnT8A) over 12 months
Time Frame: Change from baseline to 12 months
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Anti-Thymocyte Globin Plus Pegylated GCSF | Placebo
Number analyzed (Participants) | 16 | 8
nmol/L | -0.07 (0.17) | -0.10 (0.32)
Statistical Analysis 1: Comparison: Anti-Thymocyte Globin Plus Pegylated GCSF vs Placebo; Test type: Superiority or Other; p = 0.79, t-test, 2 sided; Mean Difference (Net) = 0.037, 95% CI 2-sided [-0.18 to 0.23], Standard Error of Mean 0.10

9. Secondary Outcome: Percentage of Neutrophils
Description: Change in Neutrophil Count over 12 months
Time Frame: Change from baseline to 12 months
Measure: Mean (Standard Deviation); unit: Percentage of neutrophils
Arm/Group | Anti-Thymocyte Globin Plus Pegylated GCSF | Placebo
Number analyzed (Participants) | 16 | 8
Percentage of neutrophils | 0.21 (0.69) | 0.44 (1.19)
Statistical Analysis 1: Comparison: Anti-Thymocyte Globin Plus Pegylated GCSF vs Placebo; Test type: Superiority or Other; p = 0.163, t-test, 2 sided; Median Difference (Final Values) = -7.67, 95% CI 2-sided [-18.7 to 3.35], Standard Error of Mean 5.33

10. Secondary Outcome: Change in White Blood Count (WBC) From Baseline to 12 Months
Description: Change in WBC over 12 months
Time Frame: Change from baseline to 12 months
Measure: Mean (Standard Deviation); unit: Change in percentage of WBC
Arm/Group | Anti-Thymocyte Globin Plus Pegylated GCSF | Placebo
Number analyzed (Participants) | 16 | 8
Change in percentage of WBC | -0.51 (0.81) | 0.4 (1.25)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Anti-Thymocyte Globin Plus Pegylated GCSF | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/8
Serious Adverse Events (participants affected / at risk) | 15/16 | 3/8
Other Adverse Events (participants affected / at risk) | 15/16 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-Thymocyte Globin Plus Pegylated GCSF (N=16) | Placebo (N=8)
Lymphocyte Count Decreased (Immune system disorders) | 15 (15) | 3 (5)
Serum Sickness (Immune system disorders) | 13 (13) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 14 (14) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-Thymocyte Globin Plus Pegylated GCSF (N=16) | Placebo (N=8)
Elevated Alk Phos (Endocrine disorders) | 7 (7) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 0 (0)
Chills (Immune system disorders) | 6 (6) | 1 (1)
Fatigue (General disorders) | 6 (6) | 3 (3)
Headache (General disorders) | 13 (13) | 4 (4)
Hypoglycemia (Endocrine disorders) | 12 (12) | 5 (5)
Hyponatremia (Endocrine disorders) | 3 (5) | 2 (4)
Nausea (General disorders) | 5 (8) | 0 (0)
Others (General disorders) | 15 (84) | 5 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No